CLINICAL TRIAL: NCT01295190
Title: Substitution of Propofol by Sevoflurane During Pediatric Cardiopulmonary Bypass: Effect on Metabolic Acidosis and Clinical Outcome
Brief Title: Substitution of Propofol by Sevoflurane During Pediatric Cardiopulmonary Bypass
Acronym: PRISKIKO
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Axel Fudickar, MD, University Hospital Schleswig-Holstein
Other Study IDs: Fudickar3
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Metabolic Acidosis
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Propofol: Patients receiving Propofol during cardiopulmonary bypass.
- Sevoflurane: Patients receiving sevoflurane during cardiopulmonary bypass

SUMMARY:
Propofol has been routinely used for general anesthesia during pediatric cardiopulmonary bypass at our institution without complications. However, propofol may cause propofol infusion syndrome (PRIS), a rare, but often fatal complication mainly defined by bradycardia with progress to asystolia. Metabolic acidosis is regarded as an early warning sign of PRIS. Due to the preconditioning effects of sevoflurane and its availability for cardiopulmonary bypass, propofol has recently been substituted by sevoflurane during pediatric cardiopulmonary bypass at our institution. In this study the effect of substituting propofol by sevoflurane on metabolic acidosis and outcome are examined.

DETAILED DESCRIPTION:
In this retrospective and partially prospective observational study the charts of 200 children anesthetised for pediatric heart surgery are analysed since September 2007. 100 children received propofol and up to now 80 children received sevoflurane during cardiopulmonary bypass. Blood gas analysis, laboratory results and vital parameters are compared before and after cardiopulmonary bypass for each group. Duration of intensive care treatment and time to dismission from hospital are compared between groups. Changes relative to baseline are analysed by paired t-Test with correction for multiple testing. Differences between groups are analysed by unpaired t-Test with correction for multiple testing

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for heart surgery including cardiopulmonary bypass

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children scheduled for heart surgery including cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Metabolic acidosis during cardiopulmonary bypass | 2 hours
  Changes of pH, base excess and lactate relative to baseline are analysed.

SECONDARY OUTCOMES:
Outcome parameter | 1 month
  Duration of intensive care treatment and time to dismission from hospital are compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Fudickar, Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany